CLINICAL TRIAL: NCT01342224
Title: Exploratory Trial of Immunochemoradiotherapy for Locally Advanced Pancreatic Adenocarcinoma
Brief Title: Immunochemoradiotherapy in Patients With Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Providence Health & Services (Other)
Collaborators: Providence Cancer Center, Earle A. Chiles Research Institute (Other); Robert W. Franz Cancer Research Center (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PHS 10-141B
Record Dates: First submitted 2011-04-21; First posted 2011-04-27 (Estimated); Last update posted 2018-04-12 (Actual); Status verified 2018-04

CONDITIONS: Locally Advanced Pancreatic Adenocarcinoma
Keywords: pancreatic; cancer; adenocarcinoma; vaccine
MeSH Terms: conditions — Neoplasms; Adenocarcinoma | interventions — Tadalafil; Vaccination; Gemcitabine; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- tadalafil and vaccination (Experimental): Participants receive a 4-week course of vaccination with telomerase vaccine and GM-CSF by injection, along with a cycle of gemcitabine chemotherapy (IV). This is followed by radiation and gemcitabine given twice weekly then by another dose of vaccine.
  Interventions: Biological: tadalafil and vaccination

INTERVENTIONS:
Biological: tadalafil and vaccination — Participants receive a 4-week course of vaccination with telomerase vaccine and GM-CSF by injection, along with a cycle of gemcitabine chemotherapy (IV). This is followed by radiation and gemcitabine given twice weekly then by another dose of vaccine. Four weeks after completion of chemotherapy and radiation, participants able to have surgical treatment will have surgery followed by vaccination and chemotherapy. Participants with stable or responsive disease that cannot be treated by surgery will have vaccination and chemotherapy with 2 cycles of telomerase vaccine with GM-CSF along with gemcitabine. Participants with unresectable and progressive disease after administration of vaccine, chemotherapy and radiation treatment may transition to vaccination and chemotherapy treatment.
  Other Names: tadalafil: Cialis; gemcitabine: Gemzar; telomerase vaccine: GV1001; GM-CSF: Sargramostim (Leukine)

SUMMARY:
This study will add an immunotherapy component to chemotherapy and radiation treatment in patients who have pancreatic cancer. The objective of this study is to see if the combined treatment is safe and feasible, and if a larger study is warranted.

DETAILED DESCRIPTION:
All study participants receive an initial 4 week course of intra-dermal vaccination with telomerase vaccine (GV1001) and immune adjuvant, granulocyte macrophage colony-stimulating factor (GM-CSF), along with a cycle of gemcitabine chemotherapy. This is followed by concurrent radiation therapy and low-dose intravenous (IV) gemcitabine chemotherapy given twice weekly followed by one additional dose of vaccine.

About 4 weeks (as late as 8 weeks) after chemotherapy and radiation treatment, participants with disease that can be removed by surgery will proceed to surgery. After recovery, immunochemotherapy will resume.

Participants with stable or responsive disease that is not able to be treated with surgery will proceed to immunochemotherapy.

Immunochemotherapy will consist of 2 cycles of telomerase vaccine with GM-CSF along with gemcitabine chemotherapy. Participants with disease that is not able to be treated with surgery, or that has worsened following immunochemoradiotherapy phase of treatment may continue on study with transition to immunochemotherapy phase of treatment. Tadalafil will be administered orally on a daily basis from start of therapy (Day 1) through completion of therapy with doses held only when required in the immediate perioperative period in patients who proceed to surgery.

ELIGIBILITY:
Inclusion Criteria:

Pancreatic adenocarcinoma proven by biopsy or cytology Locally advanced, unresectable disease with absence of distant metastatic disease. The presence of non-regional retroperitoneal or abdominal adenopathy is acceptable for inclusion.

OR

Borderline resectable pancreatic adenocarcinoma (any of the following):

* Tumor abutment or encasement of a short segment of hepatic artery (without evidence of tumor extension to the celiac artery) that is amenable to resection and reconstruction
* Tumor abutment of the superior mesenteric artery involving 180 degrees or less of the circumference of the artery and without encasement
* Impingement or narrowing of the superior mesenteric vein/portal vein or short-segment (< 2 cm) occlusion of the superior mesenteric vein, portal vein, or their confluence with a suitable option for vascular reconstruction
* Eastern Cooperative Oncology Group(ECOG)Performance Status 0 or 1
* Ability to give informed consent and comply with the protocol
* Women of childbearing potential must have a negative pregnancy test and must avoid becoming pregnant while on treatment. Men must avoid fathering a child while on treatment.
* Patients with a history of psychiatric illness must be judged able to understand fully the investigational nature of the study and the risks associated with the therapy.

Exclusion Criteria:

* Age < 18 years
* History of other malignancy in the past 2 years except carcinoma in situ of the cervix or bladder, or non-melanomatous skin cancer
* Previous chemotherapy or radiation therapy for pancreatic cancer or previous radiation therapy to the target field
* Clinically active autoimmune disease or active infection
* History of heart attack (within 90 days) or stroke (within 6 months), or presence of hypertension requiring change in blood pressure medications in the last 4 weeks, hypotension, uncontrolled arrhythmias, heart failure (New York Heart Association (NYHA) Functional Classification ≥ Class 2 in last 6 months), unstable angina or angina occurring during sexual activity.
* Use of "nitrates" or nitroglycerin.
* History of hereditary degenerative retinal disorders including retinitis pigmentosa.
* Chronic systemic corticosteroid use at supra-physiologic doses (prednisone > 10 mg a day or equivalent)
* Use of recreational drugs called "poppers" like amyl nitrite and butyl nitrite.
* Laboratory values (performed within 14 days prior to enrollment) as follows:

  * Neutrophil count < 1500 cells/µL
  * Hemoglobin < 9 gm/dL (patients may be transfused to establish eligibility)
  * Platelet count < 100,000 cells/µL
  * Significant coagulopathy (INR > 1.5)
  * Significant liver or renal dysfunction
* Other medical or psychiatric conditions that in the opinion of the Principal Investigator would preclude safe participation in protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Safety | 180 Days
  Adverse events will be graded no less than weekly for the first 180 days. Post-treatment long-term follow-up will occur every 12 weeks beyond day 180 for 6 visits and then every 24 weeks thereafter until progressive disease, withdrawal from study or death. For this pilot study, adverse events and efficacy measures will be personally reviewed by the principal investigator. Both hematologic and non-hematologic toxicity will be anticipated. In conjunction with the IRB, stopping the trial will be among possible measures taken if undue toxicity or inadequate outcomes are observed.

SECONDARY OUTCOMES:
Immune Response | 18 months
  In patients having surgery: Tumor tissue obtained at the time of surgery will be examined to determine the degree of macrophage and T cell infiltration. In all patients: Multiparameter flow cytometry will determine the frequency of circulating telomerase-specific memory CD8+ T cells in blood samples obtained pre- and post- treatment. Accrual is anticipate to last 10-12 months, so post treatment samples from the last patient enrolled would be available for analysis approximately 18 months after the first patient enrolled.
Tumor Response | 180 days
  Response and progression will be evaluated in this study using the international criteria proposed by the Response Evaluation Criteria in Solid Tumors (RECIST) Committee. Changes in only the largest diameter (unidimensional measurement) of the tumor lesions are used in the RECIST criteria. Tumor measurements are made 4 times during the study, the last at 180 days after study enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Crocenzi, MD, Principal Investigator — Providence Health & Services
Locations (1):
- Providence Health & Services, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Crocenzi T, Cottam B, Newell P, Wolf RF, Hansen PD, Hammill C, Solhjem MC, To YY, Greathouse A, Tormoen G, Jutric Z, Young K, Bahjat KS, Gough MJ, Crittenden MR. A hypofractionated radiation regimen avoids the lymphopenia associated with neoadjuvant chemoradiation therapy of borderline resectable and locally advanced pancreatic adenocarcinoma. J Immunother Cancer. 2016 Aug 16;4:45. doi: 10.1186/s40425-016-0149-6. eCollection 2016. PMID 27532020